CLINICAL TRIAL: NCT05436353
Title: Validity and Relaibility of Turkish Version of The Conceptualization of Pain Questionnaire
Brief Title: Turkish Version of The Conceptualization of Pain Questionnaire
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, Ph.D., Kutahya Health Sciences University
Other Study IDs: COPAQpauksbu
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain
Keywords: pain; chronic pain; attitudes and beliefs; children
MeSH Terms: conditions — Chronic Pain; Pain; Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Turkish validity and reliability — Contact with developers and formation of steering committee Translation from English to Turkish Back translation from Turkish to English Comparison of translation Review of translated versions. Reaching consensus and development of pilot version Testing in clinical setting Revision of pilot version Testing of final version

SUMMARY:
The Conceptualization of Pain Questionnaire (COPAQ), has been presented to the literature in order to evaluate the concept of pain in children and its psychometric properties. This scale, which was developed by Salvat et al., is stated as a tool that consists of a total of 15 items and is easy to administer and respond to. The total score is calculated with the correct or incorrect answers given by the children to these items, and the higher this score, the better the child's understanding of the concept of pain. Moreover; it has been shown that the scale has good fit and internal consistency. In Turkey, there is no valid and reliable scale to evaluate the concept of pain in a child with chronic pain.

The aim of this study is to create the Turkish version of "The Conceptualization of Pain Questionnaire (COPAQ)", which evaluates the concept of pain in children with chronic pain, and to question the Turkish validity and reliability of this scale.

DETAILED DESCRIPTION:
Chronic pain is a debilitating health problem often seen in children and adolescents. Although the prevalence rate varies between 11% and 38%, this rate increases with age (1). Clinical guidelines recommend that healthcare professionals help children with chronic pain understand their pain experience (2). Studies have shown that there is a relationship between the quality of the information children receive and their adaptation to and coping with pain (3). For this reason, studies in the field of pediatrics have turned to pain neuroscience education, which provides the reconceptualization of pain through education (3). Pain neuroscience education provides the basis for understanding the mechanisms of chronic pain by focusing on the biopsychosocial markers of pain (3). A pain neuroscience training protocol called 'PNE4Kids' specific to children has been introduced in the literature and it has been explained how this training should be applied to children (4). The effectiveness of the "PNE4Kids Program" has been investigated with new studies and it has been proven that it has a positive effect on the concept of pain in children and increases their knowledge of pain (5). However, there are very few scales evaluating the effectiveness of these treatments and especially the level of pain knowledge in children (6). Recently, a new scale, The Conceptualization of Pain Questionnaire (COPAQ), has been presented to the literature in order to evaluate the concept of pain in children and its psychometric properties. This scale, which was developed by Salvat et al (6), is stated as a tool that consists of a total of 15 items and is easy to administer and respond to. The total score is calculated with the correct or incorrect answers given by the children to these items, and the higher this score, the better the child's understanding of the concept of pain. Moreover; it has been shown that the scale has good fit and internal consistency (6). In our country, there is no valid and reliable scale to evaluate the concept of pain in a child with chronic pain. The aim of this study is to create the Turkish version of "The Conceptualization of Pain Questionnaire (COPAQ)", which evaluates the concept of pain in children with chronic pain, and to question the Turkish validity and reliability of this scale.

References

1. King S, Chambers CT, Huguet A, et al. The epidemiology of chronic pain in children and adolescents revisited: a systematic review. Pain 2011;152(12): 2729-2738.
2. Palermo TM, et al. "Assessment and management of children with chronic pain: A position statement from the American Pain Society. Chicago, IL: Am Pain Soc" 2012.
3. Robins H, Perron V, Heathcote LC et al. Pain neuroscience education: state of the art and application in pediatrics. Children 2016;3(4):43.
4. Pas R, Meeus M, Malfliet A, et al. Development and feasibility testing of a Pain Neuroscience Education program for children with chronic pain: Treatment protocol. Braz J Phys Ther 2018;22(3):248-253.
5. Rheel E, Ickmans K., Wauters A, et al. The effect of a pain educational video intervention upon child pain-related outcomes: A randomized controlled study. Eur J Pain 2021;25(10):2094-2111.
6. Salvat I, Adillón C, Andrés E M et al. Development of the conceptualization of pain questionnaire: A measure to study how children conceptualize pain. Int J Environ Res Public Health 2021;18(7):3821.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with FMF (Familial Mediterranean Fever) according to the "Tel Hashomer" diagnostic criteria
* Speak Turkish
* Willing to participate

Exclusion Criteria:

* The presence of another systemic disease.
* Intraarticular steroid injection or surgery in any joint in the last 3 months

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who refferred to Pamukkale University Rheumatology Clinic will be examined by one of the researchers (specialist in rheumatology) for inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
The Turkish version of Conceptualization of Pain Questionnaire (COPAQ-TR | 10 minutes
  COPAQ-TR consist of 15 items and asks respondents to respond if they believe the items/statements to be true or false, although they are allowed to respond undecided. A score of 0 is given to incorrect responses and those marked as undecided; the sum of all the correct answers gives the total score. The higher the score, the better the participant understands the concept of pain.
Turkish version ofPediatric Quality of Life Scale (PedsQL-TR) | 10 minutes
  The Pediatric Quality of Life Inventory (PedsQL) is a 23-item generic health status instrument with parent and child forms that assesses five domains of health (physical functioning, emotional functioning, psychosocial functioning, social functioning, and school functioning) in children and adolescents ages 2 to 18.
Turkish version of Child Health Assessment Scale (CHAQ-TR) | 10 minutes
  CHAQ he Childhood Health Assessment Questionnaire (CHAQ) is a disease specific health instrument that measures functional ability in daily living activities.This 30-item questionnaire is thought to have advantages over other measures of physical function due to such aspects as its multidimensionality (it assesses 8 domains of physical function).

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Başakçı ÇALIK, Prof., Study Chair — Pamukkale University
Locations (1):
- Pamukkale University Hospitals, Denizli, Turkey (Türkiye)